CLINICAL TRIAL: NCT06839196
Title: Virtual Reality Simulation and First Aid Training for Parents of Children With Special Needs on Home Accidents
Brief Title: Home Accidents Training For Parents of CWSN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: İstanbul Topkapı University (Unknown); Kocaeli University (Other)
Responsible Party: Principal Investigator, Sıla YILMAZ, Lecturer, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GAP-2024-001
Record Dates: First submitted 2025-01-28; First posted 2025-02-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Accident at Home; Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): As part of the eligibility process, participants will complete the System Usability Scale, a Likert-type questionnaire, once at the beginning of the study. Only individuals scoring in the A+ category (96th-100th percentile) will be included in the intervention phase.
  Interventions: Other: VR and first aid training

INTERVENTIONS:
Other: VR and first aid training — Intervention Stages:
  Stage 1: Descriptive Information Form and the Home Accident Awareness Questionnaire for Parents of Children with Special Needs will be administered to the parents as pre-tests.
  Stage 2: A total of 100 parents will participate in the virtual reality simulation scenarios, organized into four separate groups of 25 for implementation.
  Stage 3: Balance assessments for children will be conducted using the Children's Balance Assessment Form, the Tinetti Balance and Gait Assessment, and the Nintendo Wii Fit Balance Board.
  Stage 4: Each group of 25 participants will receive hands-on training at three different stations focusing on basic first aid and home accidents, delivered by nurses, and transfer training provided by physiotherapists.
  Stage 5: Post-tests will be administered to the parents using the Home Accident Awareness Questionnaire for Parents of Children with Special Needs.

SUMMARY:
The main objective of this project is to raise awareness and equip parents of children with special needs with the knowledge and skills necessary to prevent home accidents through virtual reality applications. Additionally, the project aims to provide parents with basic first aid training and transfer training to ensure appropriate responses in the event of an accident. It also seeks to assess the balance status of children with special needs and to identify potential fall-related risks that may lead to home accidents.

The primary research questions this project aims to address are as follows:

* What is the level of awareness among parents of children with special needs regarding home accidents?
* What is the effect of virtual reality simulation on parental awareness of home accident risks?
* How does first aid training influence parents' ability to respond to home accidents?
* What is the impact of transfer training on parents' preparedness for home accident scenarios?
* What are the balance and gait levels of children with special needs, and how might these relate to fall risk at home?

DETAILED DESCRIPTION:
As part of the eligibility process, participants will complete the System Usability Scale, a Likert-type questionnaire, once at the beginning of the study. Only individuals scoring in the A+ category (96th-100th percentile) will be included in the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* Being able to understand and speak Turkish
* Being a parent of a child with special needs
* Having a child registered at a Barrier-Free Life Application and Research Center
* Scoring in the A+ category on the System Usability Scale, with a percentile rank between 96 and 100
* Volunteering to participate in the study

Exclusion Criteria:

- Failure to meet one or more of the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Awareness of home accidents | 2 days
  The Home Accident Awareness Questionnaire for Parents of Children with Special Needs, a 28-item form developed by the researchers, will be administered twice: once before and once after the VR training program.

SECONDARY OUTCOMES:
Balance | 1 day
  The Children's Balance Assessment Form is a yes/no assessment tool developed by the researchers to evaluate the balance status of children with special needs. It will be administered once during Stage 3 of the study.
Balance | 1 day
  The Tinetti Balance and Gait Assessment will be used to evaluate balance abilities. This tool assigns scores to specific tasks, with a maximum of 16 points for the balance subscale. A higher score indicates better balance and lower risk of falling. It will be administered once during Stage 3 of the study.
Balance | 1 day
  The Nintendo Wii Fit Balance Board will be used to evaluate balance abilities through interactive tasks. It will be administered once during Stage 3 of the study.
Gait | 1 day
  The Tinetti Balance and Gait Assessment will also be used to assess gait abilities. The gait subscale has a maximum score of 28. A higher score reflects better gait performance and mobility. This assessment will be performed once during Stage 3 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Ortabağ, Prof., Study Chair — İstanbul Topkapı University; Gönül Ertunç Gülçelik, Asst. Prof., Study Director — Kocaeli University; Ebru Sever, M.Sc., Principal Investigator — Kocaeli University; Tuba Eryiğit, M.Sc., Principal Investigator — İstanbul Topkapı University; Sıla Yılmaz, M.Sc., Principal Investigator — İstanbul Medipol University

REFERENCES:
- [Derived] Ertunc Gulcelik G, Ortabag T, Yilmaz S, Sever E, Eryigit T. Virtual reality-based home accident control simulation combined with first aid training to enhance awareness in parents of children with special needs: protocol for a single-group pre-post quasi-experimental study. BMJ Open. 2025 Oct 20;15(10):e105338. doi: 10.1136/bmjopen-2025-105338. PMID 41120168